CLINICAL TRIAL: NCT03624556
Title: Pediatric Exploratory Research Study of EGCG Use and Safety (PERSEUS)
Acronym: PERSEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Instituto Hispalense de Pediatría, Sevilla, Spain (Unknown); Hospital Universitario Marqués de Valdecilla (Other); Institut Jerome Lejeune (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, Director of the Neurosciences Department in Institut Hospital d'Investigacions Mèdiques (IMIM), PharmD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PERSEUS/1
Record Dates: First submitted 2018-06-06; First posted 2018-08-10 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Down Syndrome; Fragile X Syndrome
Keywords: Down Syndrome (DS); Fragile X Syndrome (FXS); Intellectual Development Disorder (IDD); FontUp; EGCG; Epigallocatechin gallate; Dual specificity tyrosine-phosphorylation-regulated kinase 1A (Dyrk1A); Homocysteine; Dietary supplement; Green tea; IMIM; PERSEUS
MeSH Terms: conditions — Down Syndrome; Fragile X Syndrome; Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Cohort I (Down Syndrome children): Phase II Randomized, double-blind, placebo-controlled, parallel groups to evaluate safety and tolerability of EGCG in children. The experimental group will take 10mg/kg/day of FontUp (EGCG on a dietary supplement with chocolate like shake flavor, two times a day) while the placebo group will take the same product but without the EGCG in it, taken with the same posology.
  Cohort II (Fragile X syndrome children): exploratory open label study (pilot study) to assess safety and tolerability of EGCG. These patients will receive 10mg/kg/day of FontUp.
  This cohort will only be recruited in Spanish sites.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment consists in FontUp (EGCG on a dietary supplement with chocolate like shake flavor) taken dissolved in 100mL of water two times a day (breakfast and afternoon snack). The placebo treatment is the same product but without the EGCG in it, taken with the same posology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group DS and FXS (Experimental): Cohort 1: a 35 DS children group taking EGCG FontUp. Cohort 2: a 6 FXS children group taking EGCG FontUp. (Experimental open-label)
  Interventions: Dietary Supplement: EGCG FontUp
- Control group DS (Placebo Comparator): Cohort 1: a 35 DS children group taking placebo FontUp.
  Interventions: Other: Placebo FontUp

INTERVENTIONS:
Dietary Supplement: EGCG FontUp — Intake of 10mg/kg/day of EGCG, in the form of a dietary supplement (FontUp), two times a day.
  Arms: Experimental group DS and FXS
Other: Placebo FontUp — Intake of placebo, in the form of a dietary supplement (FontUp) (without EGCG), two times a day.
  Arms: Control group DS

SUMMARY:
To evaluate safety and tolerability of epigallocatechin gallate (EGCG) in children from 6 to 12 years old with Intellectual Developmental Disorders (IDD) (Down syndrome or Fragile X syndrome).

DETAILED DESCRIPTION:
This project first objective is to evaluate the safety and tolerability of the EGCG molecule (extracted form green tea) on children from 6 to 12 years old with Intellectual Development Disorder (Down syndrome and Fragile X syndrome).

The secondary objective is to evaluate the benefits of the EGCG on attention, memory, executive functions, language and adaptive behaviour of these children. Dyrk1A and homocysteine in plasma will also be quantified, using them as biomarkers of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6 to 12 years on day 1 of treatment.
* Clinical diagnosis of DS (full trisomy 21 or translocated) confirmed by chromosomal analysis (karyotyping) (Cohort I) or molecular diagnosis for FXS (mutations or premutations on the fragile mental retardation 1 gene-Fmr1 of the X chromosome) (Cohort II). A karyotype will be performed if not available in DS population. FXS molecular diagnosis will be performed if not available in FXS population.
* A body-weight under 50 kg.
* Parent or legal guardian/representative and caregiver willing to give written informed consent.
* Mental age ≥ 3 years (Brunet-Lézine scale C version, picture naming and receptive vocabulary of the WPPSI-IV)
* Study participants must have sufficient vision and hearing to participate in study evaluations. Mild hearing loss will be allowed.
* Availability of parent/caregiver to accompany the subject to clinical visits, provide information about the subject's behavior and symptoms and ensure compliance with the medication schedule.
* Subjects must be able to understand basic instructions. Naming and comprehension tasks of the WPPSI-IV will be used as an evaluation

Exclusion Criteria:

* Study participants with a current Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of any primary psychiatric diagnosis (including autism spectrum disorder). For secondary diagnoses, such as attention deficit hyperactivity disorder, depression and conduct disorder, individuals under a fixed regime of medication (a regime that does not change in the 6 weeks prior to enrollment) are allowed as long as they are considered stable and their medication does not interfere with the progression of the study.
* Personal history of infantile spasms, of epilepsy, of severe head trauma or Central Nervous System (CNS) infections (e.g. meningitis), with the exception of a single isolated febrile seizure.
* Subjects with past history of seizures from primary causes (such as West syndrome and Lennox-Gastaut syndrome) or secondary causes.
* Clinical history of moderate or severe Obstructive Sleep Apnea (OSA) as defined by Apnea-Hypopnea Index (AHI) (>15 events per hour not well controlled by positive airway pressure therapy with stable settings) for at least 3 months prior to screening visit.
* Subjects with thyroid disease that is not controlled (elevated basal Thyroid-stimulating hormone (TSH) > 10 microU/mL) by thyroid hormone respective therapy.
* Evidence of active, clinically significant, and unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
* Cardiovascular, Systolic Blood Pressure (SBP) and/or Diastolic Blood Pressure (DBP) outside the 95th percentile for age; resting heart rate above 100 bpm.
* Cardiovascular, ECG: clinically relevant ECG abnormalities at screening. Auscultation is mandatory part of cardiovascular examination.
* Clinically significant abnormalities in laboratory test results at screening unless acceptable by the investigator.
* Life-threatening illness or major surgery in the 3 months prior to the study.
* Concomitant disease or condition or any clinically significant finding at screening that could interfere with the conduct of the study, or that would, in the opinion of the investigator, could lead to an unacceptable risk to the subject in this study.
* Patients with risk factors of liver dysfunction such as previous history of liver disease, previous clinically significant hepatic abnormalities in laboratory testing, previous allergy or intolerance with liver disorders or any clinically significant abnormalities in hepatic laboratory testing at screening
* Participation in other clinical trials in the last 3 months prior to the study.
* Concomitant use of unapproved medication.
* Current intake of vitamin supplements, catechins or products containing EGCG (i.e. TEAVIGO, Mega Green Tea capsules Life Extension or Font-UP Grand Fontaine Laboratories) for at least 3 months previous to the screening.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measure : Adverse Events | From day -5 to day 252 (through study completion)
  Medical evaluations of incidence, nature, severity and causality of Adverse Events and Serious Adverse Events (SAE).
Safety Outcome Measure: Number of participants with treatment-related adverse events with supporting evidence with blood analysis: Changes in liver function | Days -5, 5, 42, 84, 126, and 168.
  The finding of an elevated alanine transaminase (ALT) or aspartate transaminase (AST) (>3xULN), elevated total bilirubin (>2xULN)
Safety Outcome Measure: Number of participants with treatment-related adverse events with supporting evidence with blood analysis: Changes in thyroid function | Days -5, 42, 84, 126, and 168.
  Elevated TSH (>10 microU/mL) or any decrease of free T4 below the lower limit of normal values (<0.8 ng/dL)
Safety Outcome Measure: Number of participants with treatment-related adverse events with supporting evidence with blood analysis: Changes in renal function | Days -15, 84, and 168
  Serum creatinine will be measured at various time points and an increase exceeding x1.5 ULN (upper limit of normal values) that is confirmed by a repeat testing within 3 days.
Safety Outcome Measure: Number of participants with treatment-related adverse events with supporting evidence with Electroencephalography (EEG): Clinical significant changes in cerebral activity | Days -15, 84, and 168
  Electroencephalogram recording to detect epileptiform abnormalities and/or seizure activity and/or pro-convulsive effects in pediatric participants, enabling a deeper understanding of the pharmacological effects of the intervention.
Safety Outcome Measure: Measure: Number of participants with treatment-related adverse events with supporting evidence with Electrocardiogram: Clinical significant changes in QTcF | Days -56 and 168
  A QTcF (Fridericia's correction) value (mean of the three measurements) exceeding 500 ms when confirmed in repeat measurement within 15-30 minutes will be recorded as SAE.
  A QTcF value exceeding a change from screening (mean of three time-matched measurements) of 60 ms when confirmed in repeat measurement within 15-30 minutes will be recorded as SAE.
Safety Outcome Measure: Measure: Number of participants with treatment-related adverse events with supporting evidence with Echocardiogram: Clinical significant changes in size of the chambers of the heart. | Days -56 and 168
  Doppler echocardiogram is used to look at how blood flows through the heart chambers, heart valves, and blood vessels. The movement of the blood reflects sound waves to a transducer. The ultrasound computer then measures the direction and speed of the blood flowing through heart and blood vessels.
Safety Outcome Measure: Measure: Number of participants with treatment-related adverse events with supporting evidence with Echocardiogram: Clinical significant changes in pumping function of the heart. | Days -56 and 168
  This measure is known as an ejection fraction or EF.

SECONDARY OUTCOMES:
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Expressive language | Days -15, 168 and 252
  Assessed by Picture Naming (PN) (WPPSI-IV). It is a verbal Comprehension subtest. It has 24 items. The child should name the drawings shown in the stimulus book. PN measures expressive language, ability and language development. Range score 0-24. Higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Receptive language | Days -1,168 and 252
  Assessed by Receptive Vocabulary (RV)(WPPSI-IV). It is a verbal comprehension subtest. It has 31 items. The child selects the picture that best represents the word the examiner reads aloud. RV measures receptive language ability and language development. Range score 0-40. Higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Memory and Learning | Days -1,168 and 252
  Assessed by Sentence Repetition (NEPSY-II): This subtest is designed to assess the ability to repeat sentences of increasing complexity and length. The child is read a series of sentences and asked to recall each sentence immediately after it is presented. Range score 0-34. Higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Working Memory (WM) | Days -1,168 and 252
  Assessed by Picture memory (WPPSI-IV). This subtest measures visual WM. It has 35 items. The child views a stimulus page of pictures for a specified time and then selects these pictures from options on a response page, for which a set of stimuli is viewed and then recognized from among a set of responses. Range score 0-35. Higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Verbal Fluency (VF) | Days -1,168 and 252
  Subjects are asked to generate as many words as possible in 1 minute belonging to the category of "animals". No range score. A higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in inhibition behavior | Days -1,168 and 252
  Assessed by Cats & Dogs Test. 16 pictures presented on a single strip of card (two trials with two conditions, control and experimental-inhibition). Measures of task accuracy in the experimental inhibition trial (total number of correct responses, range score 0-16) and total time performance (in seconds) were included in the analyses.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in mental flexibility | Days -1,84,168 and 252
  Assessed by Dimensional Change Card Sort (DCCS). Sort a series of bivalent test cards, according to one dimension(colour) or another(shape). Range score 0-24, higher score is better outcome.
Cognitive Outcome Measure : IDD-CHILD Battery. Cognitive changes in Visual-spatial Process | Days -1,168 and 252
  Assessed by Blocks Design(WPPSI-IV). It is a visual spatial subtest which has 17 items. It measures ability to analyze and synthesize abstract visual stimuli. Range score 0-34, higher score is better outcome.
Functional Outcome Measure : IDD-CHILD Vineland Adaptive Behavior Scales Scale Parent/Caregiver Interview Form, Second Edition (VABS-II)(Vineland™-II survey version) | Days -1,168 and 252
  Changes in adaptive behavior
  * A. Communication domain: Sum of A1+A2+A3. Range Score 0-198
  * A1. Receptive subdomain: Range Score 0-40
  * A2. Expressive subdomain: Range Score 0-108
  * A3. Written subdomain: Range Score 0-50
  * B. Daily living skills domain: Sum of B1+B2+B3. Range Score 0-109
  * B1. Personal subdomain: Range Score 0-82
  * B2. Domestic subdomain: Range Score 0-48
  * B3. Community subdomain: Range Score 0-88
  * C. Socialization domain: Sum of C1+C2+C3. Range Score 0-180
  * C1. Interpersonal relationships subdomain: Range Score 0-64
  * C2. Play and leisure time subdomain: Range Score 0-62
  * C3. Coping skills subdomain: Range Score 0-60
  * Total score: Sum of A+B+C. Range Score 0-576
  For all measures: a higher score is a better outcome

OTHER OUTCOMES:
Exploratory Outcome: Efficacy Biomarkers analysis in plasma | Baseline, months 3 and 6
  Dyrk1A and homocysteine (markers of efficacy); and Catechins and EGC concentrations (EGCG metabolites).
Exploratory Outcome: Blood folate concentration | Months -1, 3 and 6
  Exploratory biomarkers: determination of folate in blood samples
Exploratory Outcome Targeted metabolomics | Months -1, 3 and 6
  In the PERSEUS project spot urine samples will be collected to further evaluate the metabolome of subjects with Down syndrome, seeking biomarkers of treatment efficacy or those differentiating responders and non-responders. Analysis will be focused in the biosynthesis and metabolism of neurotransmitters, the kynurenine pathway and the hypothalamic-hypophyseal-adrenal axis.
Exploratory Outcome: Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P) | Baseline, months 6 and 9
  Evaluating changes in executive performance. BRIEF-P is a widely used caregiver questionnaire of everyday skills reflective of abilities in the executive domain. It generates a range of scales, including scales specific to working memory and inhibitory control.Raw scores and T-scores will be derived for the following scales: inhibit, shift, emotional control, initiate, working memory, plan/organize, organization of materials and monitor.
Exploratory Outcome: Observed Memory Questionnaire Parent Form (OMQ-PF) | Baseline, months 6 and 9
  Evaluating changes in memory performance. OMQ-PF is a 27-item questionnaire designed to ascertain parental perceptions about their child's memory function. All items are rated on a 5-point Likert (from 1- Strongly agree to 5-Strongly disagree OR 1- Never to 5- Always).
Exploratory Outcome: Paediatric Quality of Life Inventory (PedsQL) | Baseline, months 6 and 9
  Evaluating Quality of life.
  The PedsQL measurement model was designed to integrate the merits of generic and disease-specific instruments to evaluate quality of life. Three modules will be used:
  1. cognitive functioning scale module. Range score 0-100
  2. generic core module. Range score 0-100
  3. family impact module. Range score 0-100 For all measures: a higher score is a better outcome
Exploratory Outcome: Children's Sleep habits questionnaire (CSHQ) | Baseline, months 6 and 9
  Rebound effects after discontinuation of treatment measures: evaluating changes sleep disturbances.
  CSHQ is a 22-item parent-report questionnaire that encompasses eight domains:
  1. bedtime resistance. Range score 0-36
  2. sleep behavior. Range score 0-24
  3. night waking. Range score 0-8
  4. morning wake up. 0-16 For all items except item 19, a higher score is a better outcome
Exploratory Outcome: Aberrant Behavior Checklist (ABC) | Baseline, months 6 and 9
  Rebound effects after discontinuation of treatment measures: evaluating changes in disrupting behaviors.
  The ABC-C is a 58-item rating scale used to assess maladaptive behaviors across five original dimensions or subscales (Items are evaluated on a four-point Liker scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree)).
  1. Irritability. Range score 0-45
  2. Hyperactivity. Range score 0-48
  3. Lethargy/Withdrawal. Range score 0-21
  4. Stereotypy. Range score 0-48
  5. Inappropriate Speech. Range score 0-12 For all measures: a higher score is a worst outcome
Exploratory Outcome: Mediterranean Diet Quality Index for children and adolescents (KidMed Questionnaire) | Baseline, months 6 and 9
  KIDMED index includes 16 questions based on the principles of the Mediterranean diet, where higher scores indicate greater adherence to healthy diet. Range score -4 -16.
Exploratory Outcome: Changes in Cognitive composite Z-score | Baseline, months 6 and 9
  This variable will be created by computing the sum of the Z-scores from tests that make up IDD-CHILD battery described in secondary outcome measures. No range score. A higher score is better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- IMIM (Institut Hospital del Mar d'Investigacions Mèdiques), Barcelona, Spain

REFERENCES:
- [Background] Nagle DG, Ferreira D, Zhou YD. Epigallocatechin-3-gallate (EGCG): chemical and biomedical perspectives. Phytochemistry. 2006 Sep;67(17):1849-55. doi: 10.1016/j.phytochem.2006.06.020. Epub 2006 Jul 31. PMID 16876833
- [Background] Megarbane A, Ravel A, Mircher C, Sturtz F, Grattau Y, Rethore MO, Delabar JM, Mobley WC. The 50th anniversary of the discovery of trisomy 21: the past, present, and future of research and treatment of Down syndrome. Genet Med. 2009 Sep;11(9):611-6. doi: 10.1097/GIM.0b013e3181b2e34c. PMID 19636252
- [Background] Khoshnood B, Greenlees R, Loane M, Dolk H; EUROCAT Project Management Committee; EUROCAT Working Group. Paper 2: EUROCAT public health indicators for congenital anomalies in Europe. Birth Defects Res A Clin Mol Teratol. 2011 Mar;91 Suppl 1(Suppl 1):S16-22. doi: 10.1002/bdra.20776. Epub 2011 Mar 4. PMID 21381186
- [Background] Vicari S, Carlesimo GA. Short-term memory deficits are not uniform in Down and Williams syndromes. Neuropsychol Rev. 2006 Jun;16(2):87-94. doi: 10.1007/s11065-006-9008-4. Epub 2006 Aug 9. PMID 16967345
- [Background] Ronan A, Fagan K, Christie L, Conroy J, Nowak NJ, Turner G. Familial 4.3 Mb duplication of 21q22 sheds new light on the Down syndrome critical region. J Med Genet. 2007 Jul;44(7):448-51. doi: 10.1136/jmg.2006.047373. Epub 2007 Jan 19. PMID 17237124
- [Background] Dowjat WK, Adayev T, Kuchna I, Nowicki K, Palminiello S, Hwang YW, Wegiel J. Trisomy-driven overexpression of DYRK1A kinase in the brain of subjects with Down syndrome. Neurosci Lett. 2007 Feb 8;413(1):77-81. doi: 10.1016/j.neulet.2006.11.026. Epub 2006 Dec 4. PMID 17145134
- [Background] Altafaj X, Dierssen M, Baamonde C, Marti E, Visa J, Guimera J, Oset M, Gonzalez JR, Florez J, Fillat C, Estivill X. Neurodevelopmental delay, motor abnormalities and cognitive deficits in transgenic mice overexpressing Dyrk1A (minibrain), a murine model of Down's syndrome. Hum Mol Genet. 2001 Sep 1;10(18):1915-23. doi: 10.1093/hmg/10.18.1915. PMID 11555628
- [Background] Belichenko PV, Kleschevnikov AM, Salehi A, Epstein CJ, Mobley WC. Synaptic and cognitive abnormalities in mouse models of Down syndrome: exploring genotype-phenotype relationships. J Comp Neurol. 2007 Oct 1;504(4):329-45. doi: 10.1002/cne.21433. PMID 17663443
- [Background] Dierssen M. Down syndrome: the brain in trisomic mode. Nat Rev Neurosci. 2012 Dec;13(12):844-58. doi: 10.1038/nrn3314. PMID 23165261
- [Background] Ji J, Lee H, Argiropoulos B, Dorrani N, Mann J, Martinez-Agosto JA, Gomez-Ospina N, Gallant N, Bernstein JA, Hudgins L, Slattery L, Isidor B, Le Caignec C, David A, Obersztyn E, Wisniowiecka-Kowalnik B, Fox M, Deignan JL, Vilain E, Hendricks E, Horton Harr M, Noon SE, Jackson JR, Wilkens A, Mirzaa G, Salamon N, Abramson J, Zackai EH, Krantz I, Innes AM, Nelson SF, Grody WW, Quintero-Rivera F. DYRK1A haploinsufficiency causes a new recognizable syndrome with microcephaly, intellectual disability, speech impairment, and distinct facies. Eur J Hum Genet. 2015 Nov;23(11):1473-81. doi: 10.1038/ejhg.2015.71. Epub 2015 May 6. PMID 25944381
- [Background] Benavides-Piccione R, Dierssen M, Ballesteros-Yanez I, Martinez de Lagran M, Arbones ML, Fotaki V, DeFelipe J, Elston GN. Alterations in the phenotype of neocortical pyramidal cells in the Dyrk1A+/- mouse. Neurobiol Dis. 2005 Oct;20(1):115-22. doi: 10.1016/j.nbd.2005.02.004. PMID 16137572
- [Background] Pujol J, del Hoyo L, Blanco-Hinojo L, de Sola S, Macia D, Martinez-Vilavella G, Amor M, Deus J, Rodriguez J, Farre M, Dierssen M, de la Torre R. Anomalous brain functional connectivity contributing to poor adaptive behavior in Down syndrome. Cortex. 2015 Mar;64:148-56. doi: 10.1016/j.cortex.2014.10.012. Epub 2014 Oct 28. PMID 25461715
- [Background] de Sola S, de la Torre R, Sanchez-Benavides G, Benejam B, Cuenca-Royo A, Del Hoyo L, Rodriguez J, Catuara-Solarz S, Sanchez-Gutierrez J, Duenas-Espin I, Hernandez G, Pena-Casanova J, Langohr K, Videla S, Blehaut H, Farre M, Dierssen M; TESDAD Study Group. A new cognitive evaluation battery for Down syndrome and its relevance for clinical trials. Front Psychol. 2015 Jun 4;6:708. doi: 10.3389/fpsyg.2015.00708. eCollection 2015. PMID 26089807
- [Background] Ruiz-Mejias M, Martinez de Lagran M, Mattia M, Castano-Prat P, Perez-Mendez L, Ciria-Suarez L, Gener T, Sancristobal B, Garcia-Ojalvo J, Gruart A, Delgado-Garcia JM, Sanchez-Vives MV, Dierssen M. Overexpression of Dyrk1A, a Down Syndrome Candidate, Decreases Excitability and Impairs Gamma Oscillations in the Prefrontal Cortex. J Neurosci. 2016 Mar 30;36(13):3648-59. doi: 10.1523/JNEUROSCI.2517-15.2016. PMID 27030752
- [Background] Ruben K, Wurzlbauer A, Walte A, Sippl W, Bracher F, Becker W. Selectivity Profiling and Biological Activity of Novel beta-Carbolines as Potent and Selective DYRK1 Kinase Inhibitors. PLoS One. 2015 Jul 20;10(7):e0132453. doi: 10.1371/journal.pone.0132453. eCollection 2015. PMID 26192590
- [Background] Glasson EJ, Sullivan SG, Hussain R, Petterson BA, Montgomery PD, Bittles AH. The changing survival profile of people with Down's syndrome: implications for genetic counselling. Clin Genet. 2002 Nov;62(5):390-3. doi: 10.1034/j.1399-0004.2002.620506.x. PMID 12431254
- [Background] Martinez-Cue C, Martinez P, Rueda N, Vidal R, Garcia S, Vidal V, Corrales A, Montero JA, Pazos A, Florez J, Gasser R, Thomas AW, Honer M, Knoflach F, Trejo JL, Wettstein JG, Hernandez MC. Reducing GABAA alpha5 receptor-mediated inhibition rescues functional and neuromorphological deficits in a mouse model of down syndrome. J Neurosci. 2013 Feb 27;33(9):3953-66. doi: 10.1523/JNEUROSCI.1203-12.2013. PMID 23447605
- [Background] Pons-Espinal M, Martinez de Lagran M, Dierssen M. Environmental enrichment rescues DYRK1A activity and hippocampal adult neurogenesis in TgDyrk1A. Neurobiol Dis. 2013 Dec;60:18-31. doi: 10.1016/j.nbd.2013.08.008. Epub 2013 Aug 20. PMID 23969234
- [Background] Altafaj X, Martin ED, Ortiz-Abalia J, Valderrama A, Lao-Peregrin C, Dierssen M, Fillat C. Normalization of Dyrk1A expression by AAV2/1-shDyrk1A attenuates hippocampal-dependent defects in the Ts65Dn mouse model of Down syndrome. Neurobiol Dis. 2013 Apr;52:117-27. doi: 10.1016/j.nbd.2012.11.017. Epub 2012 Dec 5. PMID 23220201
- [Background] Guedj F, Sebrie C, Rivals I, Ledru A, Paly E, Bizot JC, Smith D, Rubin E, Gillet B, Arbones M, Delabar JM. Green tea polyphenols rescue of brain defects induced by overexpression of DYRK1A. PLoS One. 2009;4(2):e4606. doi: 10.1371/journal.pone.0004606. Epub 2009 Feb 26. PMID 19242551